CLINICAL TRIAL: NCT04814927
Title: The UMPALA Study: A Clinical Study to Assess the Impact of Contraceptives on the Cervico-Vaginal Mucosa
Brief Title: Impact of Contraceptives on Cervico-Vaginal Mucosa
Acronym: UMPALA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: CONRAD (Other); Kenya Medical Research Institute (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CONRAD D20-149
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Mucosal Inflammation; Contraceptive; Complications, Intrauterine
Keywords: Contraception; Reproductive health; Copper IUD; Etonogestrel implant; DMPA sub-cutaneous; Levonorgestrel IUS
MeSH Terms: conditions — Mucositis | interventions — Intrauterine Devices, Copper; etonogestrel; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: Participants at each site will receive one of four marketed, approved contraceptive products for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Copper IUD (Active Comparator): The copper IUD contains approximately 176 mg of copper wire wrapped around a vertical stem. It is FDA approved for pregnancy prevention for 10 years.
  Interventions: Drug: Copper IUD
- Etonogestrel Implant (Active Comparator): The ETG implant is a single, radiopaque, rod shaped implant containing 68 mg of etonogestrel. It is FDA approved for pregnancy prevention for 3 years.
  Interventions: Drug: Etonogestrel implant
- Levonorgestrel IUS (Active Comparator): The LNG IUS contains approximately 52 mg. of LNG. It is FDA approved for pregnancy prevention for 5 - 6 years.
  Interventions: Drug: Levonorgestrel IUS
- DMPA Sub-cutaneous (Active Comparator): DMPA contains 104 mg of medroxyprogesterone acetate in 0.65 mL of fluid, administered by subcutaneous injection in the abdominal fat, thigh or skin over the deltoid muscle. It is FDA approved for pregnancy prevention for 14 weeks.
  Interventions: Drug: DMPA Sub-cutaneous

INTERVENTIONS:
Drug: Copper IUD — Participants randomized to Copper IUD will receive Paragard IUD at Visit 2.
  Other Names: Paragard
  Arms: Copper IUD
Drug: Etonogestrel implant — Participants randomized to ETG implant will receive the implant at Visit 2.
  Other Names: Nexplanon; Implanon
  Arms: Etonogestrel Implant
Drug: Levonorgestrel IUS — Participants randomized to LNG intrauterine system will receive the IUS at Visit 2.
  Other Names: Mirena; Liletta
  Arms: Levonorgestrel IUS
Drug: DMPA Sub-cutaneous — Participants randomized to DMPA SC will receive the injection at Visit 2.
  Other Names: Subcutaneous depot medroxyprogesterone acetate
  Arms: DMPA Sub-cutaneous

SUMMARY:
UMPALA is a research study to look at the effect of four different, approved contraceptives on the cervical and vaginal tissues as well as on factors in the blood. Participants will have a baseline examination then receive one of four approved, marketed contraceptive products. Cervico-vaginal assessments will take place 4 weeks after contraceptive initiation and 3 months after to assess changes in mucosal safety after use of various contraceptive products in young, healthy, HIV uninfected women.

DETAILED DESCRIPTION:
This clinical study will complete approximately 12 healthy, non-pregnant, HIV-uninfected women aged 18-50 years per contraceptive arm, who are at low risk for sexually transmitted infections (STIs) at two clinical sites, for a total of approximately 96 completed participants. The study will examine changes from baseline, pre-contraceptive dosing to post contraceptive dosing of cervico-vaginal mucosal safety and adverse events.

Participants at each site will be randomized (1:1:1:1) to one of four, marketed, approved contraceptive dosing forms: Levonorgestrel (LNG) 52 mg. Intrauterine System (IUS), Copper Intrauterine Device (IUD), etonogestrel (ETG, Nexplanon, Implanon) contraceptive implant, or DMPA SC contraceptive injection.

Enrollment is expected to take approximately 8 months and each participant is expected to complete the study within 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive
* In general good health without any significant systemic disease and with an intact uterus and cervix.
* History of Pap smears and follow-up consistent with standard, local clinical practice or willing to undergo a Pap smear at Visit 1
* Willing to give voluntary consent and sign an informed consent form
* Willing and able to comply with protocol requirements, including accepting randomization to study contraceptive products
* If currently on a contraceptive product, willing to go off products and use condoms for birth control for a specified time
* If in a relationship, must be with a partner who is not known to be HIV positive and has no know risk of sexually transmitted infections (STIs)

Exclusion Criteria:

* Positive pregnancy test or plans to become pregnant during the course of the study
* Currently exclusively breastfeeding or planning to exclusively breastfeed during the course of the study
* Less than six weeks from a delivery of an infant greater than 20 weeks gestation
* Use of DMPA in the past 4 months
* Clinical signs and symptoms of menopause
* Current WHO or CDC medical eligibility criteria level 3 or 4 for any contraceptive product to which a participant could receive at the clinical site
* History of sensitivity/allergy to any component of the study product, topical anesthetic, or to both silver nitrate and Monsel's solution
* Current infection with Trichomonas vaginalis (TV), Neisseria gonorrhea (NG), Chlamydia trachomatis (CT)
* Current positive test for HIV
* History of a pulmonary embolus or deep vein thrombosis
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc)
* Known blood disorder, eg. von Willebrands disease, that could lead to prolonged or continuous bleeding with biopsy
* Chronic use systemic corticosteroids, antibiotics, antimycobacterials, anticoagulants or other drugs known to prolong bleeding and/or promote clotting, antifungals, or antivirals or antiretrovirals.
* Current or anticipated chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen for the duration of the study
* Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
* Abnormal finding on laboratory or physical examination or a social or medical condition in which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of the data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with changes to mucosal function | 4 weeks and 3 months after product use
  Evaluate mucosal factors and microbiome changes from baseline associated with mucosal function and reproductive health, including vaginal glycogen, pH, lactic acid, soluble markers and immune cells.
Number of participants with changes to mucosal health | 4 weeks and 3 months after product use
  Evaluate mucosal factors and microbiome changes from baseline associated with mucosal function and reproductive health, including vaginal glycogen, pH, lactic acid, soluble markers and immune cells.

SECONDARY OUTCOMES:
Number of participants with systemic inflammation | 4 weeks and 3 months after product use
  Evaluate changes from baseline in systemic factors associated with reproductive health, including C reactive protein and hormone concentrations.

OTHER OUTCOMES:
Mucosal susceptibility to pathogens | 4 weeks and 3 months after product use
  Model mucosal susceptibility to STIs ex vivo at baseline and after contraceptive use

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Thurman, Principal Investigator — Eastern Virginia Medical School, CONRAD
Locations (2):
- Eastern Virginia Medical School, Norfolk, Virginia, United States
- KEMRI, Thika, Central, Kenya

IPD SHARING:
Plan to Share IPD: No